CLINICAL TRIAL: NCT02905578
Title: A Phase II Trial of Pharmacological Ascorbate, Gemcitabine, and Nab-Paclitaxel for Metastatic Pancreatic Cancer (PACMAN 2.1)
Brief Title: A Phase 2 Trial of High-dose Ascorbate for Pancreatic Cancer (PACMAN 2.1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph J. Cullen (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Holden Comprehensive Cancer Center (Other); McGuff Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph J. Cullen, Professor, Department of Surgery, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201801759; 3P30CA086862 (NIH); 5U01CA140206 (NIH); P01CA217797 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Neoplasms; Cancer of Pancreas; Cancer of the Pancreas; Neoplasms, Pancreatic; Pancreas Cancer; Pancreas Neoplasms; Adenocarcinoma
Keywords: Ascorbate; Vitamin C; Pharmacological ascorbate; Pharmacologic ascorbate; Ascorbic Acid; gemcitabine; nab-paclitaxel; Gemzar; Abraxane
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbate group (Experimental): Each cycle is 4 calendar weeks
  Gemcitabine: 1000 mg/m2, once weekly for 3 weeks nab-paclitaxel: 125 mg/m2, once weekly for 3 weeks Pharmacological ascorbate: 75 grams, three times weekly for 4 weeks
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: Pharmacological ascorbate
- Control (Active Comparator): Each cycle is 4 calendar weeks
  Gemcitabine: 1000 mg/m2, once weekly for 3 weeks nab-paclitaxel: 125 mg/m2, once weekly for 3 weeks Each cycle has 1 rest week
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Administered intravenously the same day as nab-paclitaxel and ascorbate Administered after nab-paclitaxel and before ascorbate
  * given for 3 weeks out of the 4 week cycle
  * standard dose reductions are used
  * up to 2 cycles are administered before standard of care CT scan
  * decision to continue therapy is based disease response to therapy as measured from the CT scan
  * treatment continues until disease progression is identified
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: nab-paclitaxel — Administered intravenously the same day as nab-paclitaxel and ascorbate Administered after before gemcitabine and ascorbate
  * given for 3 weeks out of the 4 week cycle
  * standard dose reductions are used
  * up to 2 cycles are administered before standard of care CT scan
  * decision to continue therapy is based disease response to therapy as measured from the CT scan
  * treatment continues until disease progression is identified
  Other Names: Abraxane
Drug: Pharmacological ascorbate — Administered intravenously the same day as nab-paclitaxel and gemcitabine Administered after nab-paclitaxel and gemcitabine
  * given 3 times weekly
  * given for 4 weeks out of the 4 week cycle
  * no dose reductions are used
  * up to 2 cycles are administered before standard of care CT scan
  * decision to continue therapy is based disease response to therapy as measured from the CT scan
  * treatment continues until disease progression is identified
  Other Names: Ascorbate; Vitamin C; Ascorbic acid
  Arms: Ascorbate group

SUMMARY:
This clinical trial adds high-dose ascorbate (vitamin C) to the standard of care regimen for metastatic pancreatic adenocarcinoma (a type of pancreatic cancer). Subjects are randomized between a control group (standard treatment) and an intervention group (pharmacologic ascorbate in addition to the standard treatment).

DETAILED DESCRIPTION:
One of the standard treatments for metastatic pancreatic adenocarcinoma is nab-paclitaxel with gemcitabine. This standard therapy administers chemotherapy once per week for three weeks; patients then get a 'rest week' to complete the cycle (1 cycle = 4 weeks).

This study adds 75 grams of ascorbate (vitamin C, sometimes called pharamcological ascorbate because the dose is so high) to standard therapy. The ascorbate is administered intravenously - through a vein in the arm.

Participants in the control group will:

* receive gemcitabine and nab-paclitaxel chemotherapy, which is standard for their cancer.
* undergo imaging which is standard for their cancer and therapy. This can include CT scans, PET scans, and X-rays

Participants in the intervention group will:

* receive 75 grams of ascorbate 3 times per calendar week for each week of the chemotherapy cycle.
* undergo imaging which is standard for their cancer and therapy. This can include CT scans, PET scans, and X-rays
* provide blood samples to determine the biological effects, if any, the ascorbate has on the body during therapy.

This active therapy portion lasts until the disease progresses and a new treatment needs to be adopted - this can be months to years. If disease progresses, participants go back to standard follow-up for their caner and the new/additional therapy their doctors prescribe.

However, it is very important we remain in contact with participants; they will have life-long follow-up for this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis (cell samples, biopsy, brushing, surgical sample) of adenocarcinoma of the pancreas. Cancer from the Ampullae of Vater is also eligible. The tissue sample can be from a metastatic location, like a lymph node.
* Metastatic or node positive disease
* One cancer site, that did not receive radiation therapy, that is at least 1 cm in size when looking at it by CT scan (CAT scan)
* Recommended to receive gemcitabine and nab-paclitaxel
* Failed initial therapy or be ineligible for definitive curative therapy (e.g., surgical excision, radiation therapy)
* A platelet count of at least 100,000 cells per mL
* A creatinine level of less than 1 1/2 times the upper limit of normal for the local lab test, or, a creatinine clearance of at least 60 mL/(min*1.73m2)
* Not pregnant
* Commit to using birth control during the study (all participants)

Exclusion Criteria:

* Prior chemotherapy to treat the metastatic disease
* Other therapy (including radiation) within the past 4 weeks
* Side effects from prior therapies that are still deemed moderate to severe by a physician
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients actively receiving insulin or who are currently recommended to receive insulin by a doctor
* Patients requiring daily finger-stick blood glucose measurements
* Patients who are on the following drugs and cannot have a substitution (or who decline the substitution):

  * warfarin
  * flecainide
  * methadone
  * amphetamines
  * quinidine
  * chlorpropamide
* An active cancer, other than the pancreatic cancer, that requires treatment.
* Enrolled in another therapeutic clinical trial
* Uncontrolled, intercurrent illness
* HIV positive individuals undergoing therapy due to known drug:drug interaction between antiretroviral drugs and high-dose ascorbate therapy
* Women who are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Overall survival | Every 2 months for up to 20 years post-treatment
  Time, measured in months, from the start of chemotherapy (C1D1) to death from any cause.

SECONDARY OUTCOMES:
Tumor Response | Every 2 months for up to 10 years
  Determine the objective response rate of the disease, assessed every 2 months using CT or MRI, and evaluated/defined using the RECIST criteria (v1.1). Results are provided in nominal categories (CR, PR, SD, PD) as per RECIST.
Progression free survival | Every 2 months for up to 10 years
  Time, measured in days, it takes disease to progress, where disease progression is defined by the RECIST criteria (v1.1). Timeframe is from radiation day 1 to date of disease progression.
Adverse event frequency and categorization | Monthly through 30 days after end of treatment.
  Categorize and quantify adverse events using the Common Terminology Criteria for Adverse Events (CTCAE v4). Assessments will be monthly through 30 days past the end of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Cullen, MD, FACS, Study Director — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared per consent document, governing Federal regulations and institutional policies, and only after a signed sharing agreement between the sponsor and the requesting investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Initial requests can be submitted to the sponsor Joseph Cullen, MD, FACS at any time with a description as to the information needed.
Access Criteria: A signed usage and confidentiality agreement must be executed prior to data sharing.

REFERENCES:
- [Background] Doskey CM, Buranasudja V, Wagner BA, Wilkes JG, Du J, Cullen JJ, Buettner GR. Tumor cells have decreased ability to metabolize H2O2: Implications for pharmacological ascorbate in cancer therapy. Redox Biol. 2016 Dec;10:274-284. doi: 10.1016/j.redox.2016.10.010. Epub 2016 Oct 28. PMID 27833040
- [Background] Schoenfeld JD, Sibenaller ZA, Mapuskar KA, Wagner BA, Cramer-Morales KL, Furqan M, Sandhu S, Carlisle TL, Smith MC, Abu Hejleh T, Berg DJ, Zhang J, Keech J, Parekh KR, Bhatia S, Monga V, Bodeker KL, Ahmann L, Vollstedt S, Brown H, Shanahan Kauffman EP, Schall ME, Hohl RJ, Clamon GH, Greenlee JD, Howard MA, Schultz MK, Smith BJ, Riley DP, Domann FE, Cullen JJ, Buettner GR, Buatti JM, Spitz DR, Allen BG. O2⋅- and H2O2-Mediated Disruption of Fe Metabolism Causes the Differential Susceptibility of NSCLC and GBM Cancer Cells to Pharmacological Ascorbate. Cancer Cell. 2017 Apr 10;31(4):487-500.e8. doi: 10.1016/j.ccell.2017.02.018. Epub 2017 Mar 30. PMID 28366679
- [Derived] Bodeker KL, Smith BJ, Berg DJ, Chandrasekharan C, Sharif S, Fei N, Vollstedt S, Brown H, Chandler M, Lorack A, McMichael S, Wulfekuhle J, Wagner BA, Buettner GR, Allen BG, Caster JM, Dion B, Kamgar M, Buatti JM, Cullen JJ. A randomized trial of pharmacological ascorbate, gemcitabine, and nab-paclitaxel for metastatic pancreatic cancer. Redox Biol. 2024 Nov;77:103375. doi: 10.1016/j.redox.2024.103375. Epub 2024 Oct 2. PMID 39369582